CLINICAL TRIAL: NCT00000895
Title: Pathogenesis of MAC Disease in Advanced HIV-1-Infected Subjects and the Impact of Highly-Active Antiretroviral Treatment (HAART) on Immune Functions Relevant for MAC and Other Opportunistic Infections
Brief Title: A Study to Learn More About MAC Disease and the Use of Anti-HIV Drugs in Patients With Advanced HIV Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 341; 11312 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Mycobacterium Avium-intracellulare Infection; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Mycobacterium avium-intracellulare Infection; HIV-1; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; Mycobacterium avium Complex; Bacteremia; Nevirapine; HIV Protease Inhibitors; Risk Factors; RNA, Viral; Reverse Transcriptase Inhibitors; Nelfinavir
MeSH Terms: conditions — Mycobacterium avium-intracellulare Infection; HIV Infections; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome; Bacteremia | interventions — Nelfinavir; Nevirapine; Azithromycin

INTERVENTIONS:
Drug: Nelfinavir mesylate
Drug: Nevirapine
Drug: Azithromycin

SUMMARY:
The purpose of this study is to determine if infection with Mycobacterium avium complex (MAC) occurs in other parts of the body before it is found in the blood. This study also evaluates the relationships between the amount of HIV in the blood, immune system functions, and the presence of MAC infection.

HIV-positive patients are at risk for MAC infection because their immune systems have been weakened by HIV. It is hoped that aggressive treatment with anti-HIV drugs may improve their immune systems enough to prevent against MAC.

DETAILED DESCRIPTION:
The intent of this study is to define more precisely the natural history and immunopathogenesis of MAC disease in the HIV-infected population. It is suggested that MAC disease in AIDS patients results both from specific immunologic deficiencies caused by HIV infection of the host and as a result of specific mycobacterial virulence properties. Therefore, aggressive antiretroviral drug treatment of HIV-infected patients at risk for DMAC due to specific immune deficiencies will improve these immune functions in such a manner as to resist DMAC.

A total of 85 patients will be stratified at baseline into one of three groups:

Group I - 40 patients at high risk for MAC infection are neither followed beyond baseline nor receive study treatment.

Group II - 15 patients with DMAC, i.e., newly diagnosed MAC-bacteremic patients with no more than 72 hours prior treatment for MAC, receive individualized regimen of HAART for 48 weeks: nelfinavir (NEV), nevirapine (NVP), and nucleoside reverse transcriptase inhibitor(s) as per primary physician. Patients are evaluated through clinical, microbiologic, and virologic assessments, and intensive immunologic evaluations at Weeks 12, 24, and 48.

Group III - 30 asymptomatic HIV-infected patients are further stratified (15 patients/stratum) by CD4 count (less than or equal to 50 cells/mm3 or 100-250 cells/mm3). Patients in Group III follow the same HAART regimen and evaluations as Group II patients and continue evaluations for up to 48 weeks, if an acceptable response is found within 12 weeks of entry. Patients in Stratum 1 of Group III receive MAC prophylaxis with azithromycin once weekly with follow-up evaluations as in Group II. Patients in Group III that have a positive MAC blood or bone marrow culture at any time during the study will, from that point on, follow the same schedule of evaluations as patients in Group II.

[AS PER AMENDMENT 11/3/98: Up to 100 evaluable patients will now be studied. Group 2 is now modified to include up to an additional 15 evaluable patients with known MAC bacteremia and less than or equal to 7 days prior MAC treatment who are unable to commit to long-term follow-up (Group 2b); these patients will undergo only baseline evaluations. Group 2a consists of 15 evaluable patients with known MAC bacteremia and less than or equal to 7 days of prior MAC treatment who are willing and able to enter the follow-up phase.]

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are HIV-positive.
* Have a CD4 count under 50 cells/mm3 or between 100 and 250 cells/mm3 within 30 days of study entry.
* Have at least one symptom (e.g., fever, diarrhea, or weight loss) suggestive of MAC infection.
* Have MAC infection with 7 days or less of MAC treatment.
* Have an HIV blood level greater than 10,000 copies/ml within 30 days of study entry.
* Are 18 years of age or older.

Exclusion Criteria

You will not be eligible for this study if you:

* Have any active infection (except for MAC in Group 2 patients) or any cancer.
* Are unable to follow an acceptable anti-HIV drug regimen (Groups 2 and 3).
* Are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85
Dates: Study Completion 2001-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rob Roy MacGregor, Study Chair; David Perlman, Study Chair
Locations (26):
- United States (26):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Univ of Southern California / LA County USC Med Ctr, Los Angeles, California
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - Stanford Univ Med Ctr, Stanford, California
  - Howard Univ, Washington D.C., District of Columbia
  - Univ of Miami School of Medicine, Miami, Florida
  - Emory Univ, Atlanta, Georgia
  - Northwestern Univ Med School, Chicago, Illinois
  - Cook County Hosp, Chicago, Illinois
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Division of Inf Diseases/ Indiana Univ Hosp, Indianapolis, Indiana
  - SUNY / Erie County Med Ctr at Buffalo, Buffalo, New York
  - Beth Israel Med Ctr, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - St Vincent's Hosp / Mem Sloan-Kettering Cancer Ctr, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - Univ of Cincinnati, Cincinnati, Ohio
  - Case Western Reserve Univ, Cleveland, Ohio
  - Ohio State Univ Hosp Clinic, Columbus, Ohio
  - Univ of Pennsylvania at Philadelphia, Philadelphia, Pennsylvania
  - Julio Arroyo, West Columbia, South Carolina
  - Univ of Texas Southwestern Med Ctr of Dallas, Dallas, Texas
  - Univ of Texas, Southwestern Med Ctr of Dallas, Dallas, Texas
  - Univ of Texas Galveston, Galveston, Texas
  - Univ of Washington, Seattle, Washington

REFERENCES:
- [Result] MacGregor RR, Hafner R, Wu JW, Murphy RL, Perlman DC, Bermudez LE, Inderlied CB, Picker LJ, Wallis RS, Andersen JW, Mahon LF, Koletar SL, Peterson DM; ACTG Protocol 341 Team. Clinical, microbiological, and immunological characteristics in HIV-infected subjects at risk for disseminated Mycobacterium avium complex disease: an AACTG study. AIDS Res Hum Retroviruses. 2005 Aug;21(8):689-95. doi: 10.1089/aid.2005.21.689. PMID 16131307